CLINICAL TRIAL: NCT03766997
Title: A Randomized Controlled Study on the Effectiveness of Local Injection Combined With Topical Steroids vs. Topical Steroids Mono-therapy in the Treatment of Idiopathic Granulomatous Mastitis
Brief Title: Local Steroid Treatment for Idiopathic Granulomatous Mastitis (LSTIGM)
Acronym: LSTIGM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-breast-IGM
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Granulomatous Mastitis
Keywords: Granulomatous Mastitis; local injection; topical steroids
MeSH Terms: conditions — Granulomatous Mastitis | interventions — hydrocortisone-17-butyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local injection (Experimental): Compound betamethasone injection (Each injection contains betamethasone dipropionate at 5 mg for betamethasone and betamethasone sodium phosphate at 2 mg for betamethasone) was local injected to the breast by the patient once a week for one to four times followed by Hydrocortisone butyrate cream(0.1%) topical use twice a day until the termination of treatment.
  Interventions: Drug: Compound Betamethasone Injection; Drug: Hydrocortisone Butyrate 0.1% Cream
- topical (Active Comparator): Hydrocortisone butyrate 0.1% cream was applied to the breast by the patient twice a day until the termination of treatment.
  Interventions: Drug: Hydrocortisone Butyrate 0.1% Cream

INTERVENTIONS:
Drug: Compound Betamethasone Injection — local injection
  Arms: local injection
Drug: Hydrocortisone Butyrate 0.1% Cream — topical use

SUMMARY:
This study evaluates the clinical response rate of local steroids in the treatment of idiopathic granulomatous mastitis in female adults. Half of the participants will receive local injection combined with topical steroids and the other half will receive topical steroids mono-therapy.

DETAILED DESCRIPTION:
Idiopathic granulomatous mastitis (IGM) is a rare benign inflammatory breast disease of unknown etiology.Clinical presentation of IGM can be variable. Some findings may be confused with breast malignancy.

Although IGM as a disease has been known for nearly four decades, no treatment consensus has been reached because of its rarity. Surgical treatment, antibiotics, oral steroids, topical steroids, immunosuppression (methotrexate, mycophenolate mofetil) and close follow up have all been reported to be effective.

Currently,surgical treatment and systemic steroids treatment are most frequently employed. With the consideration of side effects of long term systemic (oral) steroid usage, topical steroids without systemic use were assessed and showed satisfactory curative effect. But there is no data concerning the use of local injection of steroids therapy on IGM.The purpose of this study is to evaluate the effectiveness of steroids local injection on the basis of topical steroids for IGM treatment.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Granulomatous Mastitis
* Require non-surgical treatment

Exclusion Criteria:

* Breast Carcinoma

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
clinical response rate | six months
  The clinical response is categorized into ''completely healed,'' ''inadequately healed,'' ''stable,'' ''worsened,'' or ''relapsed'' if the lesions had once healed but symptoms returned.

SECONDARY OUTCOMES:
granulomatous mastitis recurrence | two years
  IGM relapses in the Ipsilateral breast.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Sun, Master, Study Director — Peking Union Medical College Hospital
Locations (1):
- Department of Breast Surgery,Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tahmasebi S, Karami MY, Maalhagh M. Granulomatous Mastitis: Time to Introduce New Weapons. World J Surg. 2016 Nov;40(11):2827-2828. doi: 10.1007/s00268-016-3438-9. No abstract available. PMID 26920409
- [Background] Altintoprak F, Kivilcim T, Yalkin O, Uzunoglu Y, Kahyaoglu Z, Dilek ON. Topical Steroids Are Effective in the Treatment of Idiopathic Granulomatous Mastitis. World J Surg. 2015 Nov;39(11):2718-23. doi: 10.1007/s00268-015-3147-9. PMID 26148520
- [Background] Sheybani F, Naderi HR, Gharib M, Sarvghad M, Mirfeizi Z. Idiopathic granulomatous mastitis: Long-discussed but yet-to-be-known. Autoimmunity. 2016 Jun;49(4):236-9. doi: 10.3109/08916934.2016.1138221. Epub 2016 Feb 1. PMID 26829298
- [Background] Benson JR, Dumitru D. Idiopathic granulomatous mastitis: presentation, investigation and management. Future Oncol. 2016 Jun;12(11):1381-94. doi: 10.2217/fon-2015-0038. Epub 2016 Apr 12. PMID 27067146